CLINICAL TRIAL: NCT03081455
Title: A Prospective Evaluation of the Impact of a Process Engineering Intervention on Screening and Testing Outcomes for Common Hereditary Cancer Syndromes in Community-Based Obstetrics and Gynecology Settings
Brief Title: Impact of a Process Intervention on Screening and Testing Outcomes for Common Hereditary Cancer Syndromes
Status: Completed | Type: Observational
Sponsor: Myriad Genetic Laboratories, Inc. (Industry)
Collaborators: Myriad Genetics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PC-005
Record Dates: First submitted 2017-03-01; First posted 2017-03-16 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Hereditary Cancer
Keywords: Screening; Hereditary Cancer
MeSH Terms: interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women meeting guidelines for genetic testing: Women who present for an OB/GYN office visit (new patient visit, well woman visit, or problem visit) and who meet guidelines for genetic diagnostic testing will provide a blood or saliva sample for genetic diagnostic testing and complete a satisfaction survey.
  Interventions: Diagnostic Test: Diagnostic Test

INTERVENTIONS:
Diagnostic Test: Diagnostic Test — Genetic Diagnostic Testing

SUMMARY:
A prospective, non-interventional study to evaluate the impact of a process engineering intervention on screening and testing outcomes for common hereditary cancer syndromes in community-based OB/GYN settings.

DETAILED DESCRIPTION:
This is a prospective process intervention study that will compare historical pre-process intervention data to post-intervention data from study providers within participating community obstetrics and gynecology practices. This study will begin with a process intervention at the participating practices during which Myriad Genetics personnel experienced in implementation of hereditary cancer risk assessment programs will provide training to practice providers. The training will be followed by a 4-week practice period to allow for incorporation of the recommendations of the intervention process into the practice. During a subsequent 8-week Observation period, women who present for an office visit (new patient visit, well women visit, or problem visit) will be screened for common hereditary cancer syndromes following the process established during the process intervention. Patients who meet NCCN/ACOG testing guidelines will be offered genetic testing. Patients and study providers will be surveyed about their satisfaction with the hereditary cancer risk assessment process.

ELIGIBILITY:
Inclusion Criteria:

* Patient who presents for a new patient gynecologic visit, well woman exam, or problem gynecologic visit and meets guidelines (HBOC-NCCN guidelines; Lynch syndrome-SGO/ACOG guidelines) for genetic testing
* Patient who is 18 years of age or older
* Able to understand informed consent and agrees to participate

Exclusion Criteria:

* Patient who has previously undergone BRCA1/2, Lynch syndrome genetic testing, or multi-gene, pan-cancer, or panel testing
* Patient who is not pregnant
* Patient who is unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women presenting for a well woman visit, new patient visit, or problem visit at participating OB/GYN practices during the 8-week Observation Period.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-08-04 (Actual)

PRIMARY OUTCOMES:
The percentage of previously untested patients meeting guidelines who are offered genetic testing on site. | Baseline
  The percentage of previously untested patients meeting guidelines who are offered genetic testing on site.

SECONDARY OUTCOMES:
The number of previously untested patients meeting guidelines who agree to undergo genetic testing without a pre-test referral to a genetic counselor. | Baseline
  The number of previously untested patients meeting guidelines who agree to undergo genetic testing without a pre-test referral to a genetic counselor.

CONTACTS AND LOCATIONS:
Overall Officials: Rocye T. Adkins, MD, Study Director — Myriad Genetics, Inc.
Locations (2):
- United States (2):
  - Westwood Women's Health, Waterbury, Connecticut
  - Associates for Women's Medicine, Syracuse, New York

IPD SHARING:
Plan to Share IPD: Yes
Disclosed via peer-reviewed journal